CLINICAL TRIAL: NCT03141307
Title: The Effect of Electronic Informed Consent Information (EICI) on Residual Newborn Specimen Research
Acronym: EICI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Collaborators: Michigan Department of Health and Human Services (Other); Case Western Reserve University (Other); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Erin Rothwell, Ph.D., University of Utah
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 81352; 1R01HD082148 (NIH)
Record Dates: First submitted 2017-04-26; First posted 2017-05-05 (Actual); Results first posted 2019-09-20 (Actual); Last update posted 2019-10-01 (Actual); Status verified 2019-04

CONDITIONS: Neonatal Screening
Keywords: Neonatal screening; Biobank; Broad Consent

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Active Comparator): The EICI intervention group will receive an electronic interactive tool with movie clips and external links available through the tool. The movie intervention group will watch the educational consent movie and receive the standard paper-based brochure.
  Interventions: Behavioral: EICI Movie; Behavioral: EICI App
- Control (Placebo Comparator): This group will receive the standard of care currently used (paper-based brochure)
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: EICI Movie — The purpose of this intervention is to improve comprehension about broad consent for future biobank-dependent research by watching a brief video.
  Arms: Intervention
Behavioral: EICI App — The purpose of this intervention is to improve comprehension about broad consent for future biobank-dependent research by exploring an educational app.
  Arms: Intervention
Behavioral: Control — Standard of care, paper-based brochure
  Arms: Control

SUMMARY:
Obtaining adequate informed consent from potential research participants is a significant challenge for biobank-dependent research. To maintain public trust and support, it is important to establish an informed decision-making process for the collection and use of biospecimens collected within clinical settings. For the majority of all infants born in the US, residual dried blood biospecimens are generated after newborn screening is completed. Some programs choose to store these specimens for several uses including biomedical research. Identifying ways to improve comprehension about broad consent for future biobank-dependent research is a national priority. Specific Aim 1: Identify the key information items necessary to make an informed decision about broad consent for the retention and future research use of residual biospecimens. Methods include focus groups with new parents to determine key information elements relevant to consent for use of residual biospecimens within the Michigan BioTrust. Additional meetings with IRB personnel within the participating hospitals, health departments and universities will also be conducted to ascertain their expectations and requirements for the consent process. Specific Aim 2: Based on the data collected in Aim 1, create a state-of-the-art electronic informed consent information (EICI) tool for use in the clinical setting about the retention and use of residual biospecimens. The award-winning Genetic Science Learning Center will develop the professional EICI in Spanish and English. Validation of the EICI will be completed using feedback from both community and scientific advisory boards for the Michigan BioTrust. Specific Aim 3: Evaluate the EICI consent approach by comparing it to: a) traditional consent delivered on an electronic tablet; and b) the current paper-based consent approach. Both Spanish and English speaking parents (n = 630) in the state of Michigan, where informed consent is required for biobank research during postpartum clinical care, will be recruited and randomized to one of three groups. Specific Aim 4: Assess feasibility of the EICI through focus groups and interviews with birthing hospitals and Department of Community Health staff before and after the intervention.

* Hypothesis 1) Women in the Interactive technology group (Group A) and the video group (Group B) will demonstrate higher knowledge at Time 1 and Time 2 about the consent elements and the BioTrust than those who do not receive either EICI tool (Group C).
* Hypothesis 2) Women in the EICI groups (Groups A and B) will demonstrate lower decisional conflict at Time 1 and Time 2 toward biobanking than those who do not receive the EICI (Group C).
* Hypothesis 3) Women in the EICI groups (Groups A and B) will not differ significantly in their choices about biobanking and attitudes toward NBS and biobank research compared to participants who do not receive EICI tool (Group C).

DETAILED DESCRIPTION:
For the intervention, a research assistant (RA) at each hospital, with permission of the healthcare professional, will ask potential participants if they are interested in participating in this study. If they are interested, the RAs will seek verbal consent for this study at this time. The RA will inform patients that when a healthcare provider comes into their room about the BioTrust, they will have the study information for them.

Then the RAs at the labor and deliver units of the hospitals will give an iPad to the healthcare providers seeking consent for the BioTrust. The healthcare providers will be blind to the study group assignment until they enter the patient's room. When a healthcare professional enters a patients' room, she will touch the iPad to see the study group assignment. Participants will be randomized to one of three study groups and this will be programmed automatically on the iPad. If they are in Group A or B, the healthcare providers will give the iPad to the patients to watch or read the consent information. If they are in Group C (control group) the standard brochure will be given about the BioTrust. Immediately following their decision, all participants will complete a brief knowledge survey on the iPad.

This recruitment approach mirrors the current clinical encounter for the BioTrust. This current approach is as follows. After newborn screening is completed, a healthcare professional approaches the mother in the hospital and provides them with the Michigan BioTrust brochure (see appendix) and then asks for the mother to consent to allow or not allow their infants' residual DBS to be stored in the Michigan BioTrust. This consent form is a simply check for yes and no with their signature and is attached to the back of the newborn screening card. For this study, after they receive the information in any of the study groups, all participants will still be required to sign this same consent form because it is attached to the physical sample of the newborn screening blood specimens.

All participating women will complete a survey 1) immediately following the intervention/control on the electronic table (Time 1) and 2) also will be surveyed by telephone 2-4 weeks follow up (Time 2).

Drs. Rothwell, Johnson and Tarini will provide guidance for the coordination of the clinical sites, due to their extensive experience. To ensure success there will be at least weekly communication between the sites and the Project Director, Dr. Johnson and monthly among the site personnel. Drs. Botkin, Rothwell and Johnson will visit each site prior to implementation of data collection to introduce the project and discuss issues sites may have. Once the RAs have been hired at each site they will provide weekly reports of activities and recruitment to the Research team in Utah. Monthly a teleconference will be held and the Site PI's will report on activities and recruitment to the Utah research team and the other site PI. Consistency among the sites will be monitored with these reports and communication strategies. Research team coordination with communication and meetings is based on the successful accomplishment of previous research project (R01 HD058854).

ELIGIBILITY:
Inclusion criteria

* adult (> 18 years)
* English-speaking
* Recently given birth and are already being approached for participation in the Michigan BioTrust.
* Partner of woman who has recently given birth and is already being approached for participation in the Michigan BioTrust

Exclusion criteria

* Newborn baby is in the NICU
* Unable to speak English

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 711 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2018-06-15 (Actual); Study Completion 2018-06-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Erin Rothwell, PhD, Principal Investigator — University of Utah; Jeffrey Botkin, MD, Principal Investigator — University of Utah
Locations (1):
- Michigan Department of Health & Human Services, Lansing, Michigan, United States

IPD SHARING:
Plan to Share IPD: No
Individual data regarding knowledge about retention of newborn screening dried bloodspots is not useful data

REFERENCES:
- [Background] Joffe S, Cook EF, Cleary PD, Clark JW, Weeks JC. Quality of informed consent in cancer clinical trials: a cross-sectional survey. Lancet. 2001 Nov 24;358(9295):1772-7. doi: 10.1016/S0140-6736(01)06805-2. PMID 11734235
- [Background] Beskow LM, Dombeck CB, Thompson CP, Watson-Ormond JK, Weinfurt KP. Informed consent for biobanking: consensus-based guidelines for adequate comprehension. Genet Med. 2015 Mar;17(3):226-33. doi: 10.1038/gim.2014.102. Epub 2014 Aug 21. PMID 25144889
- [Background] O'Connor AM. Validation of a decisional conflict scale. Med Decis Making. 1995 Jan-Mar;15(1):25-30. doi: 10.1177/0272989X9501500105. PMID 7898294
- [Derived] Rothwell E, Johnson E, Wong B, Goldenberg A, Tarini BA, Riches N, Stark LA, Pries C, Langbo C, Langen E, Botkin J. Comparison of Video, App, and Standard Consent Processes on Decision-Making for Biospecimen Research: A Randomized Controlled Trial. J Empir Res Hum Res Ethics. 2020 Oct;15(4):252-260. doi: 10.1177/1556264620913455. Epub 2020 Apr 3. PMID 32242760

RESULTS

PARTICIPANT FLOW:
Period: In-Hospital
Arm/Group | Intervention | Control
Started | 471 | 240
Completed | 467 | 238
Not Completed | 4 | 2
Not completed — Withdrawal by Subject | 0 | 2
Not completed — Protocol Violation | 4 | 0
Period: Follow-Up
Arm/Group | Intervention | Control
Started | 467 | 238
Completed | 370 | 184
Not Completed | 97 | 54
Not completed — Lost to Follow-up | 97 | 54

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention | Control | Total
Number analyzed (Participants) | 471 | 240 | 711
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.78 (4.92) | 30.53 (4.76) | 30.03 (4.86)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 432 | 228 | 660
  Male | 39 | 12 | 51
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 25 | 10 | 35
  Not Hispanic or Latino | 433 | 225 | 658
  Unknown or Not Reported | 13 | 5 | 18
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 1 | 3
  Asian | 17 | 12 | 29
  Native Hawaiian or Other Pacific Islander | 2 | 0 | 2
  Black or African American | 48 | 23 | 71
  White | 362 | 184 | 546
  More than one race | 14 | 7 | 21
  Unknown or Not Reported | 26 | 13 | 39
Region of Enrollment [Number; unit: participants]
  United States | 471 | 240 | 711

OUTCOME MEASURES:

1. Primary Outcome: Comprehension for Biobanking at Time of Consent
Description: Questions based on the 16-item biobank checklist developed from consensus-based guidelines for adequate comprehension for biobanking (see Beskow et al. 2014). This measure assesses a person's understanding of the Michigan BioTrust program.
  Scale range: 0-1 The reported scale is derived from the number of correct answers divided by 20 for a percentage correct. Thus, a score of .6 indicates a 60% correct response rate. Higher values indicate more comprehension of the presented information. Lower values indicate less comprehension of the presented information.
Time Frame: Administered immediately after the intervention
Population: The analysis population differs from the number of participants enrolled because the initial 15 to 20 participants at each hospital were considered to be run-in participants during which the protocol was evaluated for its effectiveness at that site and adjusted as needed. Our analysis plan was written to exclude these run-in participants.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 444 | 225
score on a scale | .699 (.133) | .645 (.172)
Statistical Analysis 1: Comparison: Intervention vs Control; Test type: Equivalence — 95% margin; p < .001, t-test, 2 sided — a priori threshold for statistical significance set for p < .05

2. Secondary Outcome: Quality of Informed Consent
Description: The Quality of Informed Consent assesses how well the participant self-reports their understanding different aspects of the study he/she consented into (Joffe et al., 2001). Scores range from 1 to 5 with higher scores indicating better self-reported understanding of the elements of consent. The scale is created by taking the mean of 14 items.
Time Frame: Administered immediately after the intervention
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 442 | 222
score on a scale | 4.23 (.692) | 4.06 (.800)
Statistical Analysis 1: Comparison: Intervention vs Control; Test type: Equivalence — 95% margin; p < .05, t-test, 2 sided — a priori threshold for statistical significance set for p < .05

3. Secondary Outcome: Attitudes Survey
Description: Assesses support of the Michigan BioTrust program. This is a single item assessment. Full scale range is 1 to 4. Higher values indicate more support of the Michigan BioTrust. The scale is a likert scale: 1 = Not supportive at all, 4 = Very supportive
Time Frame: Administered at the 2-4 week follow-up
Population: The number of participants analyzed does not match the numbers in the participant flow due to missing data at the question level. Participants were not required to answer every single question on the survey.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 338 | 167
score on a scale | 3.62 (.626) | 3.57 (.662)
Statistical Analysis 1: Comparison: Intervention vs Control; Test type: Equivalence — 95% margin; p = .502, t-test, 2 sided — a priori threshold for statistical significance set for p < .05

4. Secondary Outcome: Residual Comprehension for Biobanking
Description: This is a repetition of the Comprehension for Biobanking survey assessed immediately after the intervention. The residual Comprehension for Biobanking survey assesses a person's retention of knowledge of the Michigan BioTrust program two to 4 weeks after the intervention.
  Scale range: 0-1 The reported scale is derived from the number of correct answers divided by 20 for a percentage correct. Thus, a score of .6 indicates a 60% correct response rate. Higher values indicate more comprehension of the presented information. Lower values indicate less comprehension of the presented information.
Time Frame: Administered at the 2-4 week follow-up
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 360 | 178
score on a scale | .693 (.153) | .667 (.159)
Statistical Analysis 1: Comparison: Intervention vs Control; Test type: Equivalence — 95% margin; p = .071, t-test, 2 sided — a priori threshold for statistical significance set for p < .05

5. Secondary Outcome: Residual Quality of Informed Consent
Description: Assessment of how well the participant understood different aspects of the study after a gap in time.
  The Residual Quality of Informed Consent is a repetition of the Quality of Informed Consent measure, now provided 2-4 weeks after the intervention. This measure assesses how well the participant self-reports their understanding different aspects of the study he/she consented into (Joffe et al., 2001). Scores range from 1 to 5 with higher scores indicating better self-reported understanding of the elements of consent. The scale is created by taking the mean of 14 items.
Time Frame: Administered at the 2-4 week follow-up
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 358 | 177
score on a scale | 4.14 (.779) | 4.03 (.763)
Statistical Analysis 1: Comparison: Intervention vs Control; Test type: Equivalence — 95% margin; p = .124, t-test, 2 sided — a prior threshold for statistical significance set for p < .05

6. Secondary Outcome: Residual Decisional Regret
Description: The Residual Decisional Regret measure assesses a person's feelings of regret after making a decision (in this specific case, participation in the Michigan BioTrust). Scores range from 1 to 5 with lower values indicating better outcomes due to less regret. The scale is created by taking the mean of 5 items.
Time Frame: Administered at the 2-4 week follow-up
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 356 | 176
units on a scale | 1.74 (.866) | 1.60 (.623)
Statistical Analysis 1: Comparison: Intervention vs Control; Test type: Equivalence — 95% margin; p < .05, t-test, 2 sided — a priori threshold for statistical significance set for p < .05

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Intervention | Control
All-Cause Mortality (participants affected / at risk) | 0/471 | 0/240
Serious Adverse Events (participants affected / at risk) | 0/471 | 0/240
Other Adverse Events (participants affected / at risk) | 0/471 | 0/240

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-03-06): https://cdn.clinicaltrials.gov/large-docs/07/NCT03141307/Prot_SAP_000.pdf